CLINICAL TRIAL: NCT03741972
Title: Metabolic and Hemodynamic Effects of the Inhibitors of Type 2 Sodium Glucose Co-transporters (ISGLT2) in Diabetic Patients With Heart Failure. GLUCOSUR-IC Study
Brief Title: Metabolic and Hemodynamic Effects of the Inhibitors of Type 2 Sodium Glucose Co-transporters (ISGLT2) in Diabetic Patients With Heart Failure
Acronym: GLUCOSUR-IC
Status: Completed | Type: Observational
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Principal Investigator, Antoni Bayés Genís, Chief of the Cardiology Unit, Germans Trias i Pujol Hospital
Other Study IDs: ICO-2018-03-PA-Glucosur
Record Dates: First submitted 2018-11-12; First posted 2018-11-15 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Heart Failure
Keywords: Heart failure; Diabetes; iSGLT2
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Treatment: Patients with diabetes and heart failure that are treated with iSGLT2
  Interventions: Drug: iSGTL2

INTERVENTIONS:
Drug: iSGTL2 — Treatment with empaglifozine 10 mg/day (may be also dapaglifozine 10mg/day depending on clinical trial results)

SUMMARY:
Inhibitors of the type 2 sodium-glucose co-transporter (iSGLT2) may improve the metabolic and hemodynamic profile in patients with DM2 and heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes
* HbA1c> 6.5%
* Estimated GF> 45 ml / min
* BMI: ≥25 Kg / m2
* Stable pharmacological treatment of Heart Failure in the last 3 months

Exclusion Criteria:

* Diabetes type 1 or type LADA (presence of antibodies against GAD and/or IA-2 positive)
* DM2 with C-peptide <1 ng / mL
* GEF <45 ml / min
* Recurrent urinary tract infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with type 2 diabetes and heart failure who attend a university hospital heart failure unit.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Change in cardiac biomarkers | 12 months
  Changes in cardiac biomarkers: NTproBNP, CA125 and ST2

SECONDARY OUTCOMES:
Change in quality of life: EuroQol-5D questionnaire (EuroQol five dimension questionnaire) | 12 months
  Changes in patient's quaility of life by 5Q questionnaire (EuroQol standardised, non-disease-specific instrument for health-related quality of life with 2 parts: first one score from 3-3-3-3 (worst) to 1-1-1-1 (best) and second one which a visual scale scores form 0 (worst)-100 (best). EuroQol-a new facility for the measurement of health-related quality of life. Health Policy 1990;16:199-208. El EuroQol-5D: una alternativa sencilla para la medición de la calidad de vida relacionada con la salud en atención primaria. Aten Primaria 2001; 28:425-429.)
Improvement of pulmonary congestion | 12 months
  Changes in pulmonary congestion by pulmonary echocardiography
Improve in the 6-minute walk | 12 months
  Changes in functional capacity by the 6 minute-walk

CONTACTS AND LOCATIONS:
Overall Officials: Nuria Alonso Pedrol, Principal Investigator — Germans Trias i Pujol Hospital
Locations (1):
- Germans Trias i Pujol University Hospital, Badalona, Spain

IPD SHARING:
Plan to Share IPD: Undecided